CLINICAL TRIAL: NCT01905241
Title: Use of Real Time Instrumentation (RTI) in Total Shoulder Arthroplasty: A Clinical Case Series
Brief Title: Use of Real Time Instrumentation (RTI) in Total Shoulder Arthroplasty
Acronym: RTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Joseph Iannotti, Chief of Staff, Executive Administration Florida, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-652
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-04

CONDITIONS: Anatomic Total Shoulder Arthroplasty
Keywords: Anatomic total shoulder arthroplasty; Glenoid; Patient specific information; Computer simulation; Computer assisted tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Anatomic TSA using RTI (Experimental): During Anatomic Total Shoulder Arthroplasty (TSA), the surgeon will have use of the SmartBone and the bone cement mold made from the SmartBone (the RTI) to transfer the preoperative plan for glenoid implant positioning to the patient's anatomy.
  Interventions: Device: Anatomic TSA using RTI; Procedure: Anatomic Total Shoulder Arthroplasty

INTERVENTIONS:
Device: Anatomic TSA using RTI — Anatomic Total Shoulder Arthroplasty (TSA) will be performed using the SmartBone and Real Time Instrumentation (RTI) to transfer the preoperative plan for glenoid implant positioning to the patient's anatomy.
Procedure: Anatomic Total Shoulder Arthroplasty — Anatomic Total Shoulder Arthroplasty will be performed by the two surgeons of the study as their Standard of Care. All procedures associated with the surgery will be the same with the exception of the instrumentation used to place the guide pin for placement of the glenoid implant.

SUMMARY:
Glenoid component loosening is the most common complication of total shoulder arthroplasty. Loosening is associated with malposition of the implant as well as the quality of the glenoid bone. Past studies from our research group have addressed these problems by investigating novel surgical technologies to increase the accuracy of glenoid implant placement. Over the course of multiple IRB approved clinical trials, use of our preoperative planning software in combination with patient specific instrumentation (PSI) or intelligent reusable instrumentation (IRI) has proven to more accurately place the glenoid guide pin than conventional standard of care techniques.

Continuing the investigator's work, the investigators propose a clinical case series to evaluate a new surgical instrumentation technique that combines the features of PSI with the IRI technology that investigators have termed Real Time Instrumentation (RTI). Investigators will measure implant placement with RSA and 3D CT imaging. Investigators will measure pre-operative bone quality using quantitative CT to measure trabecular bone volume and correlate these findings with bone samples removed from the glenoid and measured by microCT and mechanical testing of the bone samples. These bone samples will be obtained as part of the routine preparation of the glenoid bone for implant placement. This bone tissue is normally removed and discarded as part of the standard of care for preparation of the bone for placement of the glenoid. Investigators have performed all of the work required to define both the safety of all components of the proposed study in the completed PSI study and the ongoing IRI study. Since application to the IRB for study of the IRI technology Custom Orthopaedic Solutions has received in April 2013 FDA approval for this technology.

DETAILED DESCRIPTION:
The study will enroll 20 patients directly into the RTI group. Investigators will have two surgeons with experience in shoulder arthroplasty and the RTI and SmartBones technology. Investigators will require a minimum of five patients from any one surgeon. All patients will have the standard of care indications for an anatomic total shoulder arthroplasty and will give informed consent for both the surgery and participation in this study. Consent and enrollment will be obtained by the surgeon during a routine office evaluation. All patients will get standard of care pre operative x-rays and CT scan at least three weeks prior to surgery. Scan quality must meet study specific criteria and investigators expect that the scans will be performed at the Cleveland Clinic. The preoperative CT scan will be placed within our preoperative planning software (OrthoVis, Cleveland Clinic). The surgeon will use this software to assess the glenoid bone pathology and select the optimal implant and placement of that implant.

Patients will have standard of care indications for primary anatomic arthroplasty and be able to get a preoperative shoulder CT scan at the Cleveland Clinic or at an outside facility so long as the study includes the entire scapula and has 1 mm or thinner sections. These parameters are required for accurate preoperative planning as well as comparison with the post operative CT scans. Standard of care pre- and post-operative x-rays (AP and axillary views) will also be obtained and can be performed at the Cleveland Clinic or acquired from another health care facility. In all patients the standard x-rays and CT images provided by the radiology department will be available to the surgeon before and during the surgery.

Using the Smartbone surrogate model, the surgeon visually compares the exposed glenoid surface to the Smartbone model to ensure that the two match for size and shape. Any adjustments to the surgical site may be done by the surgeon to optimize the match between the model and the exposed glenoid surface. Prior to molding the bone cement, bone wax is wiped onto the model to ensure proper release of the cement mold. The surgeon will then mold bone cement around the pin in the Smartbone, capturing the trajectory of the pin and the unique contours of the glenoid rim. A small pin sleeve is inserted over the pin to be embedded within the cement model. Once the bone cement has cured, it is removed from the model and placed onto the patients glenoid surface. The bone morphology captured in the mold aligns the mold to the patient's anatomy. When surgeon feels that the model has good fit of the glenoid surface, he may continue with pin placement. After placement of the guide pin, the RTI mold is removed and the remainder of the procedure is completed using the implant manufacturer's equipment and standard surgical protocols. Any adjustments in guide pin position can be performed by the surgeon based upon surgical judgment. The surgeon can make any change needed and use any means or instrument that would otherwise be used for standard of care surgery to place the guide pin in any position that the surgeon believed to be best for the patient. If the pin is changed without the use of the RTI then the patient will be excluded from this study and the reasons for failure of the RTI technology to provide accurate pin placement based upon the surgeons sole determination of accuracy will be recorded and later analyzed as a failure to treat. These patients will not receive postoperative CT Scans as investigators would not be able to use the data.

A hollow core drill bit will be used to prepare the bone in a standard manner to obtain bone cores for study. Prior to implanting the glenoid component, three 1 mm tantalum beads will be inserted into the backside pegs of the component. Investigators have developed methods to place the beads in a manner that has been used by other investigators and validated in the investigators' own experience in 22 cases enrolled in the ongoing IRI clinical study. The desired implant will be placed into a holding device and using a drill guide, a 0.9 mm hole measuring 2 mm deep will be placed in each of the three peripheral pegs of the implant. A 1 mm tantalum bead (RSA biomedical, Umsa Sweden) supplied by the company will then be press fit into the component hole. The implant will then be placed in the glenoid, aligned with the previously drilled peg holes. As standard of care, these peg holes are cemented, thus locking the beads within the implant.

Using manufacturer (RSA biomedical, Umsa Sweden) provided beads and injector gun, four to five 1 mm tantalum beads will be placed in the coracoid, acromion and glenoid. Exact placement of these beads is at the discretion of the surgeon. Patient anatomy and operative exposure will guide the surgeon to the best places to inject the beads; however the surgeon will not be confined to a specific amount of beads in a specific location. The beads just need to be spread out amongst the coracoid, acromion, and glenoid to establish reference points for the RSA imaging. Prior studies looking at shoulder joint kinematics and implant position have used this methodology of bead placement with successful study related outcomes. Investigators have successfully placed bone beads in 22 patients currently treated in the ongoing IRI clinical study without any difficulty or adverse events during or after surgery.

Postoperatively, all patients will receive a CT with Metal Artifact Reduction (MAR)and RSA (if chosen) within 3 weeks of surgery. This will be a CT Scan performed with the patient's arm by the side in a supine position using metal artifact reduction techniques. In addition patients will receive a second CT scan and RSA imaging, provided they originally got RSA, performed 1 year (± 1 month) from surgery. The second CT scan will be performed with MAR techniques and with the patient in the lateral decubitus position with their arm in the overhead position, again using metal artifact reduction techniques. The second set of images, produced with a different body and arm position, also decreases metal artifact than those obtained with the arm placed by the side. This position cannot be comfortably obtained until 3- 6 months after surgery and require healing of the tissues and rehabilitation of the shoulder. Investigators have shown that in a small number of patients the glenoid component can shift in position within the first 3-6 months after surgery making the first CT Scan more accurate for implant position. The images obtained from the postoperative CT scans are placed back into the surgical software and the 3D reconstruction of the postoperative scapula with the implants is compared to the preoperative plan. Using measurement tools within the software, developed at the Cleveland Clinic, investigators will compare the position of the actual glenoid component placed in the patient with the desired position specified by the plan. The use and validation of these imaging methods to precisely measure implant position has been performed at the Cleveland Clinic in a prior IRB approved clinical trial (IRB 10-582).

Preoperatively, the high resolution quantitative CT will measure volumetric bone mineral density and the trabecular network of the glenoid. When available, this will be applied to the preoperative CT for those patients at Cleveland Clinic, Main Campus. Patients who have their preoperative CT completed at non Main Campus facilities will have the standard of care preoperative CT. This will be done at the same visit for the standard of care preoperative CT. Micro CT imaging, which creates a 3D reconstruction of the fine bone structure, in addition to microarchitecture analysis and mechanical testing, will allow assessment of the bone tissue taken from the bone core sample. Between the preoperative imaging and the bone tissue analysis, investigators will have data to properly determine the quality of the bone stock surrounding the implant. Further correlating these data with RSA and 3D CT imaging of implant movement, investigators can fully develop cause and effect of bone quality on glenoid component loosening.

The participating surgeons will be Drs. Joseph Iannotti and Eric Ricchetti. Patients may have surgery at either Cleveland Clinic main campus or at Euclid Hospital. If the procedure is performed at Euclid Hospital, post operative CT scan and RSA (if chosen), will need to be taken at main campus within 3 weeks. The patient will be made aware of this at the time of enrollment and consent.

By comparing the computer-generated preoperative plan to postoperative component placement, investigators will be looking at three outcomes. First, the overall difference in component placement between standard of care instrumentation, intelligent reusable instrument (IRB#12-997), patient specific instruments (IRB #10-582) and real time instrumentation will be compared. Secondly, investigators will compare the placement between the technologies within and between surgeons. Thirdly, investigators will evaluate the difference in implant position between technologies based on severity of pathology. The quality of the bone core sampled will be correlated to the possible loosening of the implants.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion, a primary anatomic total shoulder arthroplasty must be indicated for the patient.

Exclusion Criteria:

* Age less than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Iannotti, MD PhD, Principal Investigator — The Cleveland Clinic; Eric T Ricchetti, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Orthopaedic and Rheumatologic Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IDP with other researchers.

REFERENCES:
- [Background] Hendel MD, Bryan JA, Barsoum WK, Rodriguez EJ, Brems JJ, Evans PJ, Iannotti JP. Comparison of patient-specific instruments with standard surgical instruments in determining glenoid component position: a randomized prospective clinical trial. J Bone Joint Surg Am. 2012 Dec 5;94(23):2167-75. doi: 10.2106/JBJS.K.01209. PMID 23224387

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anatomic TSA Using RTI
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anatomic TSA Using RTI
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  >=18 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Difference in Glenoid Component Placement (Inclination and Version)
Description: The overall difference in component placement between Real Time Instrumentation, IRI (historical data) and standard of care instrumentation (historical data) and will be compared ((Inclination and Version).
Time Frame: Two weeks post surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic TSA Using RTI
Number analyzed (Participants) | 20
degrees
  Inclination | 2.0 (1.7)
  Version | 5.3 (3.7)

2. Secondary Outcome: Difference in Glenoid Component Position Within and Between Surgeons
Description: Investigators will compare the placement of the glenoid component between RTI, IRI and standard of care technologies within and between the two surgeons.
Time Frame: Two weeks post surgery
Population: Outcome measures data not collected/ no patients analyzed for this OM. A broader study including different surgeons is required to test the effectiveness of this technology.
Arm/Group | Anatomic TSA Using RTI
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect of Severity of Shoulder Pathology
Description: Investigators will evaluate the difference in glenoid component position between RTI, IRI (historical data) and standard of care (historical data) technologies based on severity of shoulder pathology.
Time Frame: Two weeks post surgery
Population: Outcome measures data not collected/ no patients analyzed for this OM.
Arm/Group | Anatomic TSA Using RTI
Number analyzed (Participants) | 0

4. Primary Outcome: Difference in Glenoid Component Placement (AP and SP)
Description: The overall difference in component placement between Real Time Instrumentation, IRI (historical data) and standard of care instrumentation (historical data) and will be compared (Anteroposterior Position and Superoinferior Position).
Time Frame: Two weeks post surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Anatomic TSA Using RTI
Number analyzed (Participants) | 20
mm
  Anteroposterior Position | 1.4 (0.9)
  Superoinferior Position | 1.1 (1.0)

ADVERSE EVENTS:
Time Frame: Approximately 1 year from the time of surgery.
Description: Adverse events include excessive bleeding, infection, fracture nerve injury or need for revision surgery during the term of this study which is expected to be approximately 1 year from the time of surgery. All-cause mortality was not monitored/assessed for this study.
Arm/Group | Anatomic TSA Using RTI
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01905241/Prot_SAP_000.pdf